CLINICAL TRIAL: NCT05581030
Title: A Single-Arm, Open-Label Phase 1b Study of Hyper-CVAD + Calaspargase Pegol in Young Adults With Newly Diagnosed Acute Lymphoblastic Leukemia
Brief Title: CalPeg for Newly Diagnosed Acute Lymphoblastic Leukemia (ALL)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-21213
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: A.L.L.
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — CVAD protocol; calaspargase pegol; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hyper-CVAD + Calaspargase pegol Treatment (Experimental): Participants will receive calaspargase pegol administered over 1 hour with each cycle of Hyper-CVAD, mini-CVD, and late intensification, beginning with Cycle 1B. Responding patients will have dose reduction of HyperCVAD for Cycles 2B-4B. Participants with CD20+ ALL will also be given Rituximab once per cycle.
  Interventions: Drug: Hyper CVAD Protocol (Standard of Care Multi-Agent Chemotherapy); Drug: Calaspargase Pegol; Drug: Rituximab

INTERVENTIONS:
Drug: Hyper CVAD Protocol (Standard of Care Multi-Agent Chemotherapy) — Hyper-CVAD consists of two combinations of drugs (courses A and B) given in an alternating fashion. The term "hyper" refers to the hyperfractionated nature of the chemotherapy, which is given in small doses, more frequently, to minimize side effects. CVAD is the acronym of the drugs in course a: cyclophosphamide, vincristine, doxorubicin and dexamethasone.
  Course A: Cyclophosphamide days 1, 2 and 3. Vincristine days 4 and 11, Doxorubicin day 4, dexamethasone days 1-4 and 11-14, Cytarabine day 7. Mesna is also given orally with cyclophosphamide, to reduce the incidence of haemorrhagic cystitis, a common side effect of cyclophosphamide. Methotrexate, an antimetabolite, may be given when necessary to get chemotherapy past the blood brain barrier.
  Course B: Methotrexate Day 1 and Cytarabine Days 2 and 3. Dosage is individualized to the patient.
Drug: Calaspargase Pegol — Calaspargase pegol 2000 IU/m^2 (capped at 3750 IU) will be administered beginning in cycle 1B of Hyper-CVAD, and will continue at this dose for the duration of the trial.
  Other Names: Asparlas; CalPeg
Drug: Rituximab — Rituximab 375mg/m^2 will be administered once per cycle for patients with CD20+ ALL.
  Other Names: Rituxan

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of the study drug, calaspargase pegol, when given with multi-agent chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Philadelphia negative B- or T-cell acute lymphoblastic leukemia, with >10% peripheral blood or bone marrow lymphoblasts at diagnosis.
* Treatment and full recovery from arm 1A of the Hyper-CVAD regimen.
* Be willing and able to provide written informed consent/assent for the trial.
* Able to adhere to the study visit schedule and other protocol requirements.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Cardiac ejection fraction ≥ 50% by echocardiography or MUGA, as measured prior to arm 1A of Hyper-CVAD.
* Serum bilirubin and creatinine < 1.5x upper limit of normal (ULN). AST and ALT must be <3x ULN.
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test at screening. A FCBP is considered when a sexually mature female: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 12 consecutive months.
* A FCBP must agree to use of two methods of highly effective non-hormonal contraception, be surgically sterile, or abstain from heterosexual activity for the course of the study through 3 monthsafter the last dose of study treatment.
* Male subjects must agree to use an adequate method of contraception starting with the first dose of study therapy through 30 days after the last dose of study therapy. Men must agree to not donate sperm during and after the study for 3 months

Exclusion Criteria:

* Induction therapy with any regimen other than Hyper-CVAD 1A.
* Diagnosis of L3 type Burkitt's lymphoma
* Clinical evidence of active central nervous system (CNS) leukemia.
* Any major surgery or radiation therapy within four weeks.
* Diagnosis of Down Syndrome.
* Any active infection requiring systemic therapy, including HIV, Hepatitis B, and/or Hepatitis C.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator (including but not limited to unstable angina, pre-existing liver disease, recurrent pancreatitis, uncontrolled diabetes, hypertriglyceridemia, pulmonary hypertension, or severeheart failure (New York Heart Association Class III-IV).
* Recurrent thrombosis, or non-central venous catheter associated thrombosis within 3 months prior to enrollment.
* Severe comorbid conditions for which life expectancy would be <6 months.
* Patients with active (uncontrolled, metastatic) second malignancies are excluded.
* Is pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 3 months after the last dose of trial treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-29 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Mortality Rate of Hyper-CVAD after first infusion of calaspargase pegol | Up to 12 months
  Mortality rate is hypothesized to be less than 10% when combining calaspargase pegol with Hyper-CVAD.

SECONDARY OUTCOMES:
Minimal Residual Disease Remission Rate | Up to 3 years
  Minimal Residual Disease (MRD) will be studied as a dichotomous endpoint using a cutoff of 1x10^4 cells/transcripts as the lower limit for residual leukemia and presented as the percentage of patients reaching this landmark as their best response. MRD assessment will be obtained with each bone marrow biopsy assessment, every 3 months in the first year following their last cycle of therapy and every 6 months in the subsequent 2 years following their last cycle.
Progression Free Survival | Up to 42 months
  Progression Free Survival defined as the time from start of treatment to the time of progression or death.
Overall Survival | Up to 42 months
  Overall Survival (OS) will be measured from the initial date of treatment to the recorded date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Bijal Shah, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-and-studies/clinical-trial-21213/